CLINICAL TRIAL: NCT01895504
Title: ColoAssist vs. Magnetic Guided Colonoscopy - a Randomized Controlled Trial
Brief Title: ColoAssist vs. MEI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sorlandet Hospital HF (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: ColoAssist
Record Dates: First submitted 2013-07-04; First posted 2013-07-10 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-03

CONDITIONS: Colorectal Cancer; Screening
Keywords: Colonoscopy; Colorectal cancer; Adenoma
MeSH Terms: conditions — Colorectal Neoplasms; Adenoma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ColoAssist (Experimental): Screening colonoscopy with a new colonoscope with gradual stiffness
  Interventions: Device: ColoAssist
- MEI (Active Comparator): Screening colonoscopy with colonoscopes compatible with and guided by MEI
  Interventions: Device: MEI

INTERVENTIONS:
Device: ColoAssist — Screening colonoscopy with the test instrument
  Other Names: FujiFilm EC-590WI4
  Arms: ColoAssist
Device: MEI — Colonoscopy with Olympus colonoscopes and MEI guidance
  Other Names: Olympus ScopeGuide
  Arms: MEI

SUMMARY:
Colonoscopy aims to investigate the entire colon by advancing the colonoscope tip from the rectum to the cecum, a process called cecal intubation. Cecal intubation may be difficult for different reasons, and features of the colonoscope and the use of imaging devices may influence the success rate. We want to compare the performance of a new colonoscope with novel features including gradual stiffness with that of a colonoscope supplied with a magnetic endoscope imaging (MEI) device. The hypothesis is that the performance of the new instrument is non-inferior to the MEI system.

DETAILED DESCRIPTION:
The recommended cecal intubation rate in colorectal cancer (CRC) screening is 95%. The MEI system allows real time monitoring of the colonoscope position within the colon and is considered to be a useful supplement to achieve cecal intubation. However, the MEI system is costly, and trial results are equivocal regarding the actual benefits. A newly designed colonoscope (ColoAssist) with gradual stiffness throughout the colonoscope shaft has been developed to improve insertability. We want to investigate if we can achieve equal performance results with the ColoAssist instrument as with the MEI system in CRC screening. The study is designed as a two-center, single-blinded, randomized, controlled non-inferiority trial.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion in an ongoing colorectal cancer screening trial (NCT 00883792)

Exclusion Criteria:

* Excluded from the ongoing screening trial (NCT 00883792)
* Inability or unwilling to provide informed consent

Ages: 55 Years to 66 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 475 (Actual)
Dates: Start 2013-04; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Cecal intubation rate | 1 hour
  The ability to reach the cecum during colonoscopy

SECONDARY OUTCOMES:
Cecal intubation time | 1 hour
  Time to reach the cecum during colonoscopy
Adenoma detection rate | 1 hour
  The proportion of participants in whom at least one adenoma is detected
Polyp detection rate | 1 hour
  The proportion of participants in whom at least one polyp i detected
Pain | 24 hours
  Participants will be asked to score discomfort or pain during and after colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Kjetil K Garborg, MD, Principal Investigator — SSHF Kristiansand, Norway; Michael Bretthauer, PhD, Study Chair — University of Oslo
Locations (2):
- Norway (2):
  - SSHF Arendal, Arendal
  - SSHF Kristiansand, Kristiansand

REFERENCES:
- [Derived] Garborg K, Wiig H, Hasund A, Matre J, Holme O, Noraberg G, Loberg M, Kalager M, Adami HO, Bretthauer M. Gradual stiffness versus magnetic imaging-guided variable stiffness colonoscopes: A randomized noninferiority trial. United European Gastroenterol J. 2017 Feb;5(1):128-133. doi: 10.1177/2050640616639162. Epub 2016 Jun 23. PMID 28405331